CLINICAL TRIAL: NCT04252716
Title: Prospective, Randomized, Multi-centre, Observer-masked, Non-inferiority Comparison of Two Cohesive Viscoelastic Solutions: VISTHESIA v Provisc
Brief Title: VISPER: Randomised Comparison of Two OVDs in Cataract Surgery
Acronym: VISPER
Status: Completed | Type: Observational
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Other Study IDs: Visth 1.5 BER-401-19
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Cataract Senile

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VISTHESIA 1.5: Ophtalmologic surgery supported by Visthesia OVD
  Interventions: Device: OVD
- ProVisc: Ophtalmologic surgery supported by Provisc OVD
  Interventions: Device: OVD

INTERVENTIONS:
Device: OVD — Intraocular administration

SUMMARY:
To investigate that VISTHESIA 1.5 is non-inferior to Provisc with regards to elevation in IOP greater than or equal to 30 mm Hg 6 ± 2 hours post-operatively as per methodology set out in EN ISO 15798:2013 (Primary Endpoint) To compare the changes in endothelial cell count and incidences of intraocular inflammation between VISTHESIA and Provisc as per methodology set out in EN ISO 15798:2013

ELIGIBILITY:
Inclusion Criteria:

1. Patients of any gender, 50 years of age or older at the time of study enrolment
2. undergoing age-related cataract removal (phacoemulsification) and IOL implantation in one eye only
3. Patient informed of the needs and visit schedule required of the Clinical Investigational Plan and who has given his/her written informed consent
4. Planned implantation of the IOL in the capsular bag

Exclusion Criteria:

1. Patients not able to / willing to give informed consent
2. Patients not able to comprehend and comply with study requirements
3. Patients scheduled for surgery to the fellow eye within 48 hrs preceding any scheduled study follow up. (Surgery date could be changed)
4. Patients not able to attend follow-up appointments for any reason
5. Patients with known hypersensitivity to anaesthetics of the amide type or hyaluronan
6. Patients with reduced corneal endothelium (e.g. Fuch's dystrophy)
7. Patients with epilepsy, impaired cardiac conduction, bradycardia, or impaired respiratory function
8. Patients being treated with tocainide for cardiac arrhythmia
9. Patients with impaired hepatic function, if the anaesthetic dose or site of application is likely to result in high blood levels
10. Mono-ophthalmic patients
11. Patients who have previously undergone cataract surgery in the contralateral eye
12. Patients with any psychosocial, or other chronic disease conditions that may affect the perception of bodily pain
13. VISTHESIA (topical and intracameral components) or ProVisc is not a suitable device for the patient for any reason
14. Patients with other pathology or condition presenting, according to the investigator opinion, a risk for the patient (to be documented in screen log)
15. Female patients who are menstruating, pregnant, breastfeeding or amenorrheic for less than 2 years at the time of surgery
16. Patients who may require the use of hyaluronidase as part of the study cataract procedure
17. Patients who may be regarded as being vulnerable (e.g. prisoners, residents of care or mental health institutions, trauma, war or disaster victims, dependent on the investigator etc.)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in need of cataract surgery
Sampling Method: Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2022-02-08 (Actual)

PRIMARY OUTCOMES:
IOP | 6-hours post-operatively
  Frequency of incidence of Intraocular Pressure greater than or equal to 30 mm Hg

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital Freiburg, Freiburg im Breisgau, Baden-Wurttemberg, Germany